CLINICAL TRIAL: NCT04902404
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of the First Pathways Game on Parent-child Interaction Quality and Children's Development for Children Aged 3-36 Months Experiencing Adversity in Calgary
Brief Title: Evaluation of the First Pathways Game on Parent-child Interactions and Development for Vulnerable Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: International Society of Psychiatric-Mental Health Nurses (Unknown)
Responsible Party: Principal Investigator, Nicole Letourneau, Professor in the Faculty of Nursing, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB21-0415
Record Dates: First submitted 2021-04-10; First posted 2021-05-26 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Internet-Based Intervention
Keywords: randomized controlled trial; digital parenting intervention; parent-child interactions; children's developmental milestones; adverse childhood experiences; vulnerable population; infants/young children; health promotion; community-based research

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Pathways Group (Experimental): Parents in the First Pathways Game group will be instructed to log into the First Pathways website daily and play First Pathways games with their child. They will receive daily reminders for the first month after randomization but will not receive reminders for the second month.
  Interventions: Other: First Pathways Game
- Wait-list Control (No Intervention): Parents in the wait-list control group will receive access to the First Pathways game after completing their final two-month study assessment.

INTERVENTIONS:
Other: First Pathways Game — The First Pathways Game is a free, online parenting education program. Parents watch short videos (approximately 30 seconds) on the First Pathways Game website to receive neuroscience knowledge and ideas for age-appropriate game ideas to play with their child. The game ideas employ common household items, such as measuring cups and paper.
  Arms: First Pathways Group

SUMMARY:
Children's brains develop quickly in the first three years of life and are particularly sensitive to their environment. Adverse experiences, such as exposure to abuse and neglect, can increase children's risk for behavioral, mental health (e.g., depression, anxiety), and developmental struggles. Fortunately, supportive, nurturing parents can help protect children from these poor health and developmental outcomes. In-person parenting programs have been shown to improve parents' interactions with their children. However, many parents struggle to access these programs due to competing life demands and accessibility barriers (e.g., lack of transportation and childcare). The First Pathways Game is a free, online tool that was created by an expert in brain development to provide parents with games and activities for playtime with their child, based on their child's age. The investigators plan to study the impact of the First Pathways Game on parent-child interactions and development of children aged 3-36 months. The investigators will recruit families in Calgary that are experiencing adversity, such as poverty and homelessness. Parent-child pairs will be randomly assigned to the (1) First Pathways group that is reminded to play the First Pathways Game daily for a month or (2) wait-list control group, to allow for comparisons. Before, immediately after, and 2 months after the month-long program, the investigators will collect information on parent-child interactions and children's development with reliable and valid tools to examine the effectiveness of the First Pathways Game. This free, online tool has the potential to empower parents in supporting their children's health and development and could be ideal for families experiencing vulnerability, due to its accessibility. If found effective, this tool could improve both short- and long-term health outcomes for children with experiences of adversity.

DETAILED DESCRIPTION:
Background and Rationale: Exposure to early adverse childhood experiences (ACEs), such as abuse and neglect, increase children's risk for detrimental health (e.g., physical, mental, behavioral) and developmental (e.g., milestones, academic) consequences. Since children's brains develop rapidly within the first few years of life, they are remarkably sensitive to ACEs, yet positive parent-child interactions can buffer the impacts of early adversities. Although numerous, efficacious in-person parenting interventions are available, barriers (e.g., transportation, childcare) limit accessibility. Recent research has shown that families are interested in accessing parenting and child development information online, and over 80% of low-income families have internet access and internet-enabled devices. Furthermore, online interventions are of particular importance during the novel coronavirus (COVID-19) pandemic when limited in-person resources are available. The First Pathways Game (www.firstpathwaysgame.com) is a free online tool aimed at improving parent-child interactions and children's development by providing parents with age-appropriate, interactive activities. The First Pathways Game was developed by neuroscientist Dr. Judy Cameron to promote parent-child interactions and children's development by sharing neuroscience knowledge and age-appropriate game ideas for parents and children to play together. A pilot study of 16 low-income families in Pittsburgh showed improved parent-child interaction scores for children at the highest risk, offering evidence of promise as a feasible intervention.

Objective: The investigators will examine the effect of the First Pathways Game on parent-child interactions and children's developmental milestones for disadvantaged (e.g., low-income) families with children aged 3-36 months in Calgary, Alberta.

Methods: The investigators will conduct a multi-center, two-arm, parallel-group, superiority randomized controlled trial with a 1:1 allocation ratio. Parent-child pairs will be recruited from Calgary agencies that provide services for families facing adversity, such as families who have experienced domestic violence and low-income families. Data collection will be facilitated by REDCap with integrated computer-aided block randomization. Both groups will be assessed at baseline, and one and two months later with observational and parent-reported questionnaire measures. Participants will be randomized to the First Pathways group or wait-list control group after the baseline data assessment is complete. Parents in the First Pathways group will receive their choice of daily reminders (e.g., phone call, email, text message) to access the First Pathways website daily for the first month and their game utilization will be tracked by their device (phone, tablet, computer) for the two-month study duration. Parent-child pairs in the wait-list control group will receive access to the First Pathways website after the final two-month assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Child is aged 3-36 months
2. Parent has a device (e.g. cellphone, laptop) to access the internet
3. Parent has internet access
4. Parent can provide informed written consent in English

Exclusion Criteria:

1. Child has a neurodevelopmental (e.g., cerebral palsy) disorder or motor or language impairment
2. Family plans to move out of Calgary and surrounding areas within two months of study enrollment
3. Parent has received Working for Kids: Building Skills Training

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Parent-Child Interaction Quality | Parent-child interactions will be measured with the Parent-Child Interaction Teaching Scale at baseline and one and two months post randomization to assess change in parent-child interaction scores over time.
  The observational Parent-Child Interaction Teaching Scale will be utilized to measure parent-child interaction quality. Parent-child interactions are assessed while parents teach their child a new skill, with 73 binary (yes, no) observational measures. The Parent-Child Interaction Teaching scale provides total scores for parent (i.e., sensitivity to cues, responsiveness to distress, social-emotional growth fostering, cognitive growth fostering) and child (i.e., clarity of cues, responsiveness to parent) behaviors. Parental scores range from 0-50, and child behaviors range from 0-23; high scores represent optimal parent-child interactions.
Parent-Child Interaction Quality | Parent-child interactions will be measured with the Simple Interactions tool at baseline and one and two months post randomization to assess change in parent-child interaction scores over time.
  The Simple Interactions tool will be utilized as a second observational measure of parent-child interactions, and data from this research will inform the convergent validity between the Simple Interactions and Parent-Child Interaction Teaching Scale. Parent-child pairs are evaluated on three outcomes: (1) parent-child mutual social and emotional connection; (2) balanced back and forth interactions called reciprocity; and (3) parental willingness to offer appropriate challenges to their child to provide them with an opportunity to grow. Parent-child pairs can receive scores ranging from 100-500 for each outcome (i.e., connection, reciprocity, opportunity to grow), with a score of 500 indicating high optimal parent-child interactions. Additionally, an overall composite score is created by averaging the connection, reciprocity, and opportunity to grow scores.

SECONDARY OUTCOMES:
Children's gross and fine motor, communication, personal-social, and problem-solving skills. | The Ages and Stages Questionnaire Third edition will be administered at baseline and one and two months post randomization to determine if children's gross motor, fine motor, communication, personal-social, and problem-solving skills change over time.
  The Ages and Stages Questionnaires Third Edition will be utilized to measure children's gross and fine motor, communication, personal-social, and problem-solving skills. This parent-reported screening tool is comprised of 21 questionnaires for children aged 1-66 months. Each developmental domain (i.e., communication, gross motor, fine motor, problem-solving, personal-social) is comprised of six questions and scores range from 0-60; children who score below an age-determined threshold for each developmental domain are considered to have a developmental concern.
Children's social-emotional development | The Ages and Stages Questionnaire Social-Emotional Second Edition will be administered at baseline and one and two months post randomization to determine if children's social-emotional development changes over time.
  The parent-reported Ages and Stages Questionnaire Social-Emotional Second edition will be utilized to measure children's social-emotional development; this tool is employed for children aged 1-72 months and is comprised of 9 questionnaires. Score ranges differ per age group as the number of items varies between questionnaires. For example, the 6-month questionnaire includes 23 items and the 18-month questionnaire includes 31 items. Per item, scores range from 0-15, with lower scores indicative of more optimal social-emotional development. Children who score above an age-specific cut-off are considered to have a social-emotional developmental concern.

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Komanchuk, BN, Principal Investigator — University of Calgary; Nicole Letourneau, PhD, Principal Investigator — University of Calgary; Judy L Cameron, PhD, Principal Investigator — University of Calgary
Locations (1):
- Community Agencies, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No